CLINICAL TRIAL: NCT00001495
Title: A Phase I Study of Irinotecan (CPT-11) Administered as a Prolonged Infusion in Adult Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960013; 96-C-0013
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Neoplasms
Keywords: Camptothecin; Cancer; Chemotherapy; Natural Products; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan (CPT-11)

SUMMARY:
This study examines a 96 hour infusion schedule of irinotecan alternating with 72 hour drug-free intervals in patients with solid tumors in order to determine the maximum tolerated dose of this regimen.

DETAILED DESCRIPTION:
Irinotecan (CPT-11) is a promising camptothecin analogue with activity in solid tumors. In Phase I studies using short intravenous infusion schedules, the predominant drug toxicities have been gastrointestinal, such as diarrhea, and myelosuppression. In animal studies, prolonged infusion schedules followed by short drug-free intervals have resulted in preservation of antitumor activity and decreased drug toxicity. Therefore, we propose to examine a 96 hour infusion schedule of irinotecan alternating with 72 hour drug-free intervals in patients with solid tumors in order to determine the maximum tolerated dose of this regimen. The duration of these treatments will be escalated in our Phase I study until patients are receiving therapy for 2 out of every 3 weeks. Standard Phase I drug toxicity and tumor response information will be monitored and the pharmacokinetics of irinotecan and its active metabolite, SN-38 will also be examined. We will also attempt to monitor the intracellular molecular effects of SN-38 therapy in blood, bone marrow, and, whenever possible, tumor tissue.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Recurrent or metastatic cancer, including lymphoma.

No leukemia.

No active CNS disease.

Refractory to all effective therapy OR No effective therapy exists.

Measurable disease not required.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Greater than 4 weeks and recovered from immunotherapy.

Chemotherapy: Greater than 4 weeks and recovered from chemotherapy.

Previous therapy with irinotecan is permitted.

Endocrine Therapy: Not specified.

Radiotherapy: Greater than 4 weeks since radiotherapy.

Surgery: Recovered from prior surgery.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0-2.

Hematopoietic: AGC greater than 1,500.

Platelets greater than 100,000.

Hepatic: Bilirubin no greater than 1.5 mg/dL.

AST no greater than 2 times normal.

Renal: Creatinine no greater than 1.5 mg/dL.

OTHER:

HIV negative.

No active infection requiring antibiotics.

No concurrent medical illness that would interfere with chemotherapy.

No pregnant or nursing women.

Adequate contraception required of fertile patients.

Imaging/exams for tumor measurement within 28 days prior to registration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1995-11; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Negoro S, Fukuoka M, Masuda N, Takada M, Kusunoki Y, Matsui K, Takifuji N, Kudoh S, Niitani H, Taguchi T. Phase I study of weekly intravenous infusions of CPT-11, a new derivative of camptothecin, in the treatment of advanced non-small-cell lung cancer. J Natl Cancer Inst. 1991 Aug 21;83(16):1164-8. doi: 10.1093/jnci/83.16.1164. PMID 1653362
- [Background] de Forni M, Bugat R, Chabot GG, Culine S, Extra JM, Gouyette A, Madelaine I, Marty ME, Mathieu-Boue A. Phase I and pharmacokinetic study of the camptothecin derivative irinotecan, administered on a weekly schedule in cancer patients. Cancer Res. 1994 Aug 15;54(16):4347-54. PMID 8044782